CLINICAL TRIAL: NCT01056757
Title: A Phase I/II Exploratory Study of Ribavirin in Metastatic Breast Cancer Expressing Elevated eIF4E
Brief Title: Treatment With Ribavirin for Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study closed because of new overlapping study with ribavirin.
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Wilson Miller, Principal Investigator, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ribavirin-003
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; ribavirin; eIF4E
MeSH Terms: conditions — Breast Neoplasms | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ribavirin (Experimental)
  Interventions: Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — 1000 mg bid, po, q28days

SUMMARY:
The purpose of this study is to learn whether oral Ribavirin is safe and effective in treating patients with metastatic breast cancer, that have high levels of eIF4E.

DETAILED DESCRIPTION:
Overexpression of eIF4E occurs in greater than 50% of BC, where it has been associated with clinical progression, angiogenesis and chemoresistance. eIF4E protein expression is not elevated in stroma or in benign tissue. A major focus in the future management of BC is to develop novel targeted therapeutics, with associated biomarkers of clinical value. It is possible that targeting a central regulator that can control multiple pathways might be more effective than targeting a single downstream molecule. In our preclinical studies, we have demonstrated that ribavirin inhibits proliferation of BC cell lines at clinically achievable concentrations by inhibiting its target, eIF4E. This trial addresses the important clinical issue of the lack of treatment for poor prognosis BC, characterized by overexpression of eIF4E. We will explore the use of eIF4E as therapeutic target and a predictive marker. We will determine whether targeting eIF4E with ribavirin, a commercially approved, inexpensive, oral therapeutic compound with a favourable toxicity profile, may present a novel treatment option for patients with aggressive, metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer at diagnosis, with metastatic disease at the time of screening, who have progressed on prior anthracycline and taxane-containing regimens.
* Willing to have a screening biopsy performed from an easily accessible lesion (ex. skin, superficial lymph node), AND must have overexpression of eIF4E in the metastatic tissue.
* Easily accessible lesion for serial biopsies (ex. skin, superficial lymph node, or other easily accessible site).
* At least 1 unidimensionally measurable lesion (based on the RECIST criteria) outside the CNS.
* ECOG 0, 1, or 2.
* Adequate recovery (excluding alopecia) from previous surgery, radiation, and chemotherapy.
* Adequate wash-out period from last therapy for breast cancer (at least 3 weeks).
* Life expectancy ≥ 12 weeks.
* Age is ≥ 18 years. There is no upper age limit since the drug can be administered orally and even considered in a palliative setting.
* Female patients of childbearing potential must have a negative serum (beta-HCG) pregnancy test within 14 days of starting protocol and must not be breastfeeding. Men and women of childbearing potential must agree to use an effective means of contraception throughout the study and for at least 6 months after completion of protocol. Post-menopausal women (defined as 12 or more consecutive months of amenorrhea, or follicle stimulating hormone (FSH) in the post-menopausal range), or surgically sterile women, do not require methods of contraception.
* Adequate renal and hepatic function: serum creatinine < 1.5 x ULN; AST or ALT < 2.5 x ULN (or < 5 x ULN if liver involvement with metastases); serum bilirubin < 1.5 x ULN.
* Adequate hematopoietic function: neutrophils ≥1.0 x 10E9/L, platelets ≥ 100 x 10E9/L.
* Provide written consent after the investigational nature, study design, risks and benefits of the study have been explained.
* Accessible for treatment and follow up.

Exclusion Criteria:

* Symptomatic brain metastases.
* Active cardiovascular disease as defined by New York Heart Association (NYHA) class III-IV categorization.
* Intercurrent illness or medical condition precluding safe administration of the planned protocol treatment or required follow-up.
* Use of any investigational drug within 4 weeks before start of study treatment or inadequate recovery from any toxic effects of such therapy.
* Female patients who are pregnant or breastfeeding.
* Concurrent treatment with other anti-cancer therapy. Bisphosphonates are allowed as long as they were started prior to screening (at least 4 weeks before study entry) and the dose does not change during study participation.
* Known infection with HIV.
* History of other malignancy in the past 5 years. Subjects who have been disease-free for 1 year or subjects with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-12; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate to therapy with daily oral ribavirin | 2 years

SECONDARY OUTCOMES:
Time to and duration of response | 1-5years
Time to relapse | 1-5 years
To determine the medical risk (safety and tolerability) that ribavirin may have on breast cancer patients as determined by laboratory tests, vital signs, and clinical adverse events. | 1-2 years
Correlation between activity of eIF4E and response | 1-2 years
Effect of ribavirin on the activity of eIF4E related pathways | 1-2 years
Evaluate pharmacokinetic parameters of ribavirin | 1-2 years
Correlate expression of eIF4E in fresh and archived tissue | 1-2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Miller, MD, PhD, Principal Investigator — Jewish General Hospital; Katherine Borden, PhD, Study Director — Université de Montréal
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kentsis A, Topisirovic I, Culjkovic B, Shao L, Borden KL. Ribavirin suppresses eIF4E-mediated oncogenic transformation by physical mimicry of the 7-methyl guanosine mRNA cap. Proc Natl Acad Sci U S A. 2004 Dec 28;101(52):18105-10. doi: 10.1073/pnas.0406927102. Epub 2004 Dec 15. PMID 15601771
- [Background] Assouline S, Culjkovic B, Cocolakis E, Rousseau C, Beslu N, Amri A, Caplan S, Leber B, Roy DC, Miller WH Jr, Borden KL. Molecular targeting of the oncogene eIF4E in acute myeloid leukemia (AML): a proof-of-principle clinical trial with ribavirin. Blood. 2009 Jul 9;114(2):257-60. doi: 10.1182/blood-2009-02-205153. Epub 2009 May 11. PMID 19433856
- [Background] Coleman LJ, Peter MB, Teall TJ, Brannan RA, Hanby AM, Honarpisheh H, Shaaban AM, Smith L, Speirs V, Verghese ET, McElwaine JN, Hughes TA. Combined analysis of eIF4E and 4E-binding protein expression predicts breast cancer survival and estimates eIF4E activity. Br J Cancer. 2009 May 5;100(9):1393-9. doi: 10.1038/sj.bjc.6605044. Epub 2009 Apr 14. PMID 19367274
- [Background] Holm N, Byrnes K, Johnson L, Abreo F, Sehon K, Alley J, Meschonat C, Md QC, Li BD. A prospective trial on initiation factor 4E (eIF4E) overexpression and cancer recurrence in node-negative breast cancer. Ann Surg Oncol. 2008 Nov;15(11):3207-15. doi: 10.1245/s10434-008-0086-9. Epub 2008 Aug 22. PMID 18719964